CLINICAL TRIAL: NCT01531426
Title: Cerebral Oxygen Saturation as Outcome Predictor in Cardiac Arrest Patients Undergoing Mild Therapeutic Hypothermia
Brief Title: Cerebral Oxygenation in Cardiac Arrest and Hypothermia
Acronym: CoCaHYp
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Principal Investigator, C. Storm, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: CoCa-01-12
Record Dates: First submitted 2012-02-06; First posted 2012-02-13 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Cardiac Arrest
Keywords: resuscitation; hypothermia; outcome
MeSH Terms: conditions — Heart Arrest; Hypothermia | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NIRS continuous monitoring
  Interventions: Device: near infrared spectroscopy (INVOS®, Covidien)

INTERVENTIONS:
Device: near infrared spectroscopy (INVOS®, Covidien) — Measurement of regional cerebral oxygen saturation with non-invasive near-infrared INVOS® (In-Vivo Optical Spectroscopy) monitor by Covidien.
  Other Names: INVOS® (In-Vivo Optical Spectroscopy); Covidien

SUMMARY:
Data indicate that neurological prognostication is difficult after cardiac arrest if mild therapeutic hypothermia is part of the post resuscitation care. Cerebral oxygenation detected by near-infrared spectroscopy, could be a new, non-invasive index marker for outcome assessment after cardiac arrest. The investigators hypothesize that cardiac arrest survivors with a continuously low cerebral oxygenation index have a poor prognosis.

DETAILED DESCRIPTION:
The measurement of cerebral oxygen saturation by a non-invasive near-infrared monitor, INVOS® (In-Vivo Optical Spectroscopy; Covidien) can detect changes in oxygen levels reflecting regional blood oxygen saturation of the brain tissue beneath the sensor. If this monitoring can add further information towards reliable prognostication after cardiac arrest is unknown so far.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years

Exclusion Criteria:

* under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after cardiac arrest
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
neurological outcome (death; CPC: 5) | participants will be followed for the duration of hospital stay, an expected average of 3-6 weeks
  Cerebral Performance Category 5: death

SECONDARY OUTCOMES:
neurological outcome CPC 1-5 | participants will be followed for the duration of hospital stay, an expected average of 3-6 weeks and a 12 month follow up will be performed
  CPC 1: Conscious and alert with normal function or only slight disability CPC 2: Conscious and alert with moderate disability CPC 3: Conscious with severe disability CPC 4: Comatose or persistent vegetative state CPC 5: death

CONTACTS AND LOCATIONS:
Overall Officials: Christian Storm, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Universitätsmedizin, Berlin, Germany